CLINICAL TRIAL: NCT05994820
Title: Implementing and Evaluating a Chatbot-based Intervention to Promote Vaccine Acceptance in Varansi, India
Brief Title: Chatbot-based Intervention to Promote Vaccine Acceptance in Varansi, India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00023512; IRB00023512 (Other: JHSPH IRB)
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Vaccine Hesitancy
Keywords: Health Communication; Chatbot; Social Networks
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Masking Description: All parties are aware of assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): These participants receive no intervention. No chatbot messaging. Usual care.
- Vaccine Campaign (Experimental): These participants will receive the Happy Baby Programme messages through a WhatsApp Chatbot. All messages will be narrowly focused on vaccine promotion.
  Interventions: Behavioral: Happy Baby Programme -Vaccine Campaign
- Vaccine++ Campaign (Experimental): These participants will receive the Happy Baby Programme messages through a WhatsApp Chatbot. All messages will promote vaccines in conjunction with other health-promotion activities (e.g. nutrition, breastfeeding, etc.).
  Interventions: Behavioral: Happy Baby Programme- Vaccine ++ Campaign

INTERVENTIONS:
Behavioral: Happy Baby Programme -Vaccine Campaign — The Happy Baby Programme is a WhatsApp based Chatbot designed to promote childhood vaccination in Hindi.
  Arms: Vaccine Campaign
Behavioral: Happy Baby Programme- Vaccine ++ Campaign — The Happy Baby Programme is a WhatsApp based Chatbot designed to promote childhood vaccination in Hindi as part of a holistic healthy baby approach that includes nutrition and sanitation.
  Arms: Vaccine++ Campaign

SUMMARY:
The goal of this clinical trial is to learn compare the efficacy Chatbot messaging directed to parents of infants and children living in unstable urban housing (UUH) in Varansi, India. The main questions it aims to answer are: 1) Can a Chatbot intervention be used to improve attitudes towards childhood vaccines? 2) Does an intervention in which vaccination is presented in the larger context of well-being improve attitudes towards vaccination?

DETAILED DESCRIPTION:
Only 2/3 of Indian infants and children are fully immunized. In communities facing unstable urban housing (UUH) vaccination rates are even lower. COVID-19 introduced new challenges for community health workers in these areas, and many do not have the capacity to promote vaccination. At the same time, the pandemic also prompted more parents and caregivers to engage with smartphones to manage the child's health. The investigators believe that a WhatsApp-based Chatbot intervention may be an effective way to promote routine childhood vaccination among caregivers without creating additional burdens on community health workers. To test this, the investigators are developing the Happy Baby Programme. This programme will be disseminated as a Chatbot through WhatsApp to parents of infants and young children living in Varanasi, in the Indian state of Uttar Pradesh. In addition to testing the overall efficacy of a Chatbot messaging platform, the investigators will compare two different Chatbot messaging designs, one featuring vaccine-only messaging and a second that positions vaccines as part of a broader set of well-being practices.

ELIGIBILITY:
Inclusion Criteria:

* Speak Hindi;
* Reside in selected UUH neighborhood of Varanasi, India;
* Identify as a caregiver of a young child (<2) OR be at least 5 months pregnant and due to giver birth during the study period;
* Child is registered with local community health workers and included on patient rosters for vaccination clinics (also known as Village Health Sanitation and Nutrition Days (VHSNDs));
* Have regular access to a phone with WhatsApp.

Exclusion Criteria:

* Only one caregiver is eligible per household
* Not meeting inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2058 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Post Intervention Vaccine Intentions | 4 months
  Vaccine intentions will be assessed through 3-Likert type questions that ask participants to respond on a five-point scale (from strongly disagree to strongly agree, where higher scores mean more higher intentions). Responses will be averaged into an index (spanning from 0 = lowest intention to 5 = highest intention to vaccinate) to signify vaccine intentions. We will assess changes in these intentions from baseline to post-intervention.
Post Intervention Vaccine Attitudes | 4 months
  Vaccine attitudes will be assessed through an 8-item scale using Likert-style questions that ask participants to respond on a five-point scale (from strongly disagree to strongly agree, where higher scores mean more positive agreement). Responses will be averaged into an index (spanning from 0 = lowest intention to 5 = highest intention to vaccinate) to signify vaccine attitudes. We will assess changes in these attitudes from baseline to post-intervention. Please note that, in this methodology, there is no need to create a binary "negative attitude" versus "positive attitude."
Post Intervention Vaccine Hesitancy | 4 months
  Vaccine Hesitancy will be assessed through a validated 10-item scale from Shapiro et al. 2017. All items utilize a Likert-type response format. that ask participants to respond on a five-point scale (from strongly disagree to strongly agree, where higher scores mean more positive agreement) answers. Responses will be averaged into an index (spanning from 0 = most hesitancy, to 5 = least least hesitancy) to signify vaccine hesitancy. We will assess changes in hesitancy from baseline to post-intervention. Please note that, in this methodology, there is no need to create a binary "hesitant" versus "not hesitant."

SECONDARY OUTCOMES:
Parental Awareness of Vaccine Services | 4 months
  Awareness will be assessed through 2 knowledge based questions on a questionnaire administered after the intervention. Responses will scored on a three-point scale: 0 = not aware; 1 = aware but does not know the date; and 2= aware and knows the date. Higher scores correspond to greater awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv N Rimal, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- D-COR (Development Corner) Consulting, Dwārka, New Delhi, India

IPD SHARING:
Plan to Share IPD: No
All participant data will be deidentified and stored on local servers (in India). American researchers will only access deidentified data for evaluation purposes.